CLINICAL TRIAL: NCT05517889
Title: Assessing the Stability and Repeatability of OCT Features in Healthy Skin: a Test-retest Study
Brief Title: Repeatability and Stability of Healthy Skin Features on OCT
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Maastricht University (Precision medicine The D-lab) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022-3219
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Optical Coherence Tomography; Artificial Intelligence; Radiomics
Keywords: Optical coherence tomography; OCT; Artificial intelligence; AI; Radiomics; Test-retest; Imaging; Dermatology; Skin
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Optical coherence tomography — Optical coherence tomography is a non-invasive scanner which generates real-time in-vivo images of the skin and its adnexal structures. Images are generated by light-interferometry.

SUMMARY:
A test-retest study on the stability and repeatability of healthy skin features on OCT

ELIGIBILITY:
Inclusion Criteria:

* At least18 years of age

Exclusion Criteria:

* Unable to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 30 healthy volunteers (colleages from the department of dermatology (MUMC+) and precision medicine (UM) will be asked to participate in this study. They must have at least three naevi.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Repeatable hand-crafted radiomics-features | Interval of 10 minutes
  The number of HRFs that are repeatable in a test-retest setting
Interclass Correlation Coefficient (ICC) | 1 month
  Intraclass Correlation Coefficient (ICC) will be used to assess the correlation and repeatability of the HRFs resulting from OCT scans. ICC will be calculated after all scans have been obtained.
  ICC will be used to rank the HRFs. This statistical test is commonly used reliability index in test re-test studies.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht UMC+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Gathered data will only be available to the prinicpal invesitgators and involved research staff (one PhD-candidate from dermatology (MUMC+), one PhD-candidate from precision medicine (UM)).